CLINICAL TRIAL: NCT04610879
Title: Randomised Factorial Design Controlled Trial Comparing Carbamazepine, Levetiracetam or Active Monitoring Combined With or Without Sleep Behaviour Intervention in Treatment Naive Children With Rolandic Epilepsy
Brief Title: Changing Agendas on Sleep, Treatment and Learning in Epilepsy
Acronym: CASTLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Following the internal pilot, the study did not meet prespecified stop/go criteria for continuation.
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); University of Liverpool (Other); Bangor University (Other); Edge Hill University (Other); Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: CASTLE; 2018-003893-29 (EudraCT Number); RP-PG-0615-20007 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2019-07-09; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Rolandic Epilepsy
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Carbamazepine; Levetiracetam; Methods

STUDY DESIGN:
Intervention Model Description: The trial is a phase IV randomised factorial design controlled trial comparing carbamazepine, levetiracetam or active monitoring combined with or without sleep behaviour intervention. We have used a factorial trial design as this approach enables the efficient simultaneous investigation of anti-epileptic drug (AED) (carbamazepine; levetiracetam; no AED) and sleep behaviour intervention (vs standard care) by including all participants in both analyses. In a factorial trial it is also possible to consider both the separate effects of each intervention and the benefits of receiving both interventions together (for example levetiracetam and sleep intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Carbamazepine plus sleep intervention (Active Comparator)
  Interventions: Drug: Carbamazepine; Behavioral: Parent based sleep (PBS) intervention
- Carbamazepine plus standard care (Active Comparator)
  Interventions: Drug: Carbamazepine
- Levetiracetam plus sleep intervention (Active Comparator)
  Interventions: Drug: Levetiracetam; Behavioral: Parent based sleep (PBS) intervention
- Levetiracetam plus standard care (Active Comparator)
  Interventions: Drug: Levetiracetam
- No AED plus sleep intervention (Active Comparator)
  Interventions: Behavioral: Parent based sleep (PBS) intervention
- No AED plus standard care (No Intervention)

INTERVENTIONS:
Drug: Carbamazepine — Treatment will be procured, prescribed and issued as per routine NHS practice. Generics can be prescribed.
  Arms: Carbamazepine plus sleep intervention; Carbamazepine plus standard care
Drug: Levetiracetam — Treatment will be procured, prescribed and issued as per routine NHS practice. Generics can be prescribed.
  Arms: Levetiracetam plus sleep intervention; Levetiracetam plus standard care
Behavioral: Parent based sleep (PBS) intervention — The PBS intervention is an e-learning package for parents/primary carers and children with epilepsy. The PBS intervention offers parents education about normal sleep, advice about sleep-promoting practices and targeted strategies parents can employ to help their children to ''learn'' an appropriate set of sleep behaviours/habits and/or to unlearn inappropriate sleep behaviours.
  Other Names: CASTLE Online Sleep Intervention (COSI)
  Arms: Carbamazepine plus sleep intervention; Levetiracetam plus sleep intervention; No AED plus sleep intervention

SUMMARY:
Rolandic epilepsy (RE) is the most common type of epilepsy. Children with RE have seizures and can often find that their learning, sleep, behaviour, self-esteem and mood are affected.

As part of standard NHS care, children diagnosed with RE may be treated with standard anti-epileptic medicines, like carbamazepine, or no medicine at all. The medicines used to treat epilepsy often slow down a child's thinking and learning. In the past, doctors believed this was an acceptable price to pay to reduce seizures. However, with RE, where the seizures usually stop in teenage years, investigators do not know if it is better to treat these children with medicines or not, especially if the medicines might have a negative effect on their learning.

A newer medicine called levetiracetam has also been found to work in children with RE and has shown less problems with thinking and learning in adults. However, it is still no known if this is also the case for children and it has not been proven which of the three options (carbamazepine, levetiracetam or no treatment) would be best for RE patients. The CASTLE study aims to find this out.

In addition, it has been found that seizures often happen when a child has had poor sleep and they often come at night or early in the morning. It has been shown that sleep can be improved through practice without the need of medicines. There are established guidelines to help toddlers go to sleep, but nothing available that helps young people with epilepsy and their parents improve their sleep quality. In the CASTLE study, a sleep training plan has been developed for children with epilepsy and the trial aims to find out whether following this sleep training plan results in less seizures than using no sleep training at all.

DETAILED DESCRIPTION:
The trial is a phase IV randomised factorial design controlled trial comparing carbamazepine, levetiracetam or active monitoring combined with or without sleep behaviour intervention. A factorial trial design has been used as this approach enables the efficient simultaneous investigation of AED (carbamazepine; levetiracetam; no AED) and sleep behaviour intervention (vs standard care) by including all participants in both analyses. In a factorial trial it is also possible to consider both the separate effects of each intervention and the benefits of receiving both interventions together (for example levetiracetam and sleep intervention).

The CASTLE trial will take place in NHS out-patient paediatric epilepsy and general paediatric clinics in the United Kingdom (UK).

Once consent has been obtained from the appropriate adult, and assent from the child if appropriate, by the delegated member of the research team the eligibility assessments will be completed, full eligibility confirmed (confirmation must be by a medically qualified doctor) and baseline data will be collected prior to randomisation.

Randomisation will be performed via a web based tool accessed by research team at site. This system is generated centrally by the Clinical Trial Research Centre (CTRC) using a computer algorithm concealed from the investigators and research teams/trial management group. In order to balance the groups, minimisation for variables believed to influence disease outcome and end points will be built into the randomisation algorithm.

Participants will be randomised to treatment with carbamazepine, levetiracetam or active monitoring. Where randomised to drug treatment, the randomised treatment should ideally begin on the day of randomisation or within 14 days of randomisation at the latest. Randomised treatment will continue for a minimum of 12 months and a maximum of 48 months. All treatments will be procured, prescribed and issued as per routine NHS practice.

Clinical data capture will be in the form of paper copies of Case Report Forms (CRFs) that will be returned as an on-going process from each centre to the CTRC. Patient/parent reported data will be collected directly on paper at each outpatient visit with the exception of CANTAB, which will be collected on iPads at the centre.

All trial documents (except raw Hospital Episode Statistics (HES) from NHS digital that will only be retained for 1 year) will be retained for 25 years from the End of Trial. The PI at each investigational centre must make arrangements to store the essential trial documents, (as defined in Essential Documents for the Conduct of a Clinical Trial (ICH E6, Guideline for Good Clinical Practice)) including the ISF, until the CTRC informs the investigator that the documents are no longer to be retained

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with RE (see International League Against Epilepsy Diagnostic Manual at https://www.epilepsydiagnosis.org/syndrome/ects-overview.html)
2. EEG showing focal sharp waves with normal background (see International League Against Epilepsy Diagnostic Manual at https://www.epilepsydiagnosis.org/syndrome/ects-eeg.html)
3. Aged ≥5 years and <13 years at the time of randomisation
4. Currently untreated with antiepileptic drugs
5. Written informed consent received from person with parental responsibility/legal representative.
6. Family have an email address and regular internet access (for online sleep intervention)
7. Parent and child are to have a good understanding of the English language

Exclusion Criteria:

1. Known contraindication to any of the trial drugs
2. Previously treated for epilepsy with antiepileptic drugs

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Time to 6-month seizure remission | Up to 48 months
  To determine if carbamazepine or levetiracetam are superior to no anti-epileptic drugs
Change from baseline to total sleep problem score as measured by the Children's Sleep Habits Questionnaire (CSHQ) | At 3 months
  To determine if a Parent-Based Sleep intervention is superior to standard care

SECONDARY OUTCOMES:
Total costs measured in Quality-Adjusted Life Years (QALYs) | At 0, 3, 12, 24, 36 and 48 months
  To estimate the cost-utility of carbamazepine, levetiracetam and PBS
Time taken from randomisation to decision by child, parent or treating physician to be withdrawn from treatment due to inadequate seizure control or unacceptable adverse reactions | At 3, 6,12, 24, 36 and 48 months
  To compare time to treatment failure due to inadequate seizure control or unacceptable adverse reactions
Time taken from randomisation to decision by child, parent or treating physician to be withdrawn from treatment due to inadequate seizure control | At 3, 6,12, 24, 36 and 48 months
  To compare time to treatment failure due to inadequate seizure control
Time taken from recruitment to decision by child, parent or treating physician to be withdrawn from trial due to unacceptable adverse reactions | At 3, 6,12, 24, 36 and 48 months
  To compare time to treatment failure due to unacceptable adverse reactions
Time to first seizure based on seizure report | At 3, 6,12, 24, 36 and 48 months
  To compare time to first seizure
Time to 12-month seizure remission based on seizure report | At 3, 6,12, 24, 36 and 48 months
  To compare time to 12-month remission from seizures
Total sleep problem score as measured by the Children's Sleep Habits Questionnaire (CSHQ) | At 12, 24, 36 and 48 months
  To determine if a Parent-Based Sleep intervention is superior to standard care
Total score in three chosen assessments delivered by the Cambridge Neuropsychological Test Automated Battery (CANTAB) | At 0, 3, 6,12, 24, 36 and 48 months
  To compare measures of cognition across the different treatment groups
Score change in Health Related Quality of Life in Children with Epilepsy - Child self-report scale (CHEQOL) | At 0, 12, 24, 36 and 48 months
  To compare Health Related Quality of Life across the different treatment groups
Total score on Strengths and Difficulties Questionnaire (SDQ) | At 0, 12, 24, 36 and 48 months
  To compare measures of children's behaviour across the different treatment groups
Records of adverse reactions | At 3, 6, 12, 24, 36 and 48 months
  To identify any adverse reactions and their rate
Score changes in Child Health Utility instrument (CHU9D) | At 0, 3, 12, 24, 36 and 48 months
  To estimate child health utilities and Quality-Adjusted Life Years (QALYs) across the different treatment groups
Score changes in EQ-5D-Y | At 0, 3, 12, 24, 36 and 48 months
  To estimate child health utilities and Quality-Adjusted Life Years (QALYs) across the different treatment groups
EQ-5D-5L score change | At 0, 3, 12, 24, 36 and 48 months
  To estimate health utilities and Quality-Adjusted Life Years (QALYs) across parents in the different treatment groups
Score changes in Parental Self-Efficacy Measure (PSAM) | At 0, 3, 12, 24, 36 and 48 months
  To compare parenting self-efficacy across the different treatment groups
Total sickness related school absences (days) | At 0, 3, 6, 12, 24, 36 and 48 months
  To compare sickness related school absences across the different treatment groups
Resource Use Questionnaire | At 3, 12, 24, 36 and 48 months
  To determine the costs to the National Health Service (NHS)
Hospital Episode Statistics (HES) Data | 48 months, measured for the participant's study duration
  To determine the costs to the National Health Service (NHS)
Patient Level Information and Costing System (PLICS) Data | 48 months, measured for the participant's study duration
  To determine the costs to the National Health Service (NHS)

OTHER OUTCOMES:
Summary of actigraphy variables (total sleep time/sleep latency/sleep efficiency) averaged over a 1-week period | 1 week actigraphy (arranged centrally via Oxford unit) at baseline, 3 and 12 months
  To determine which sleep parameters change in primary carer and child dyads in different treatment groups

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London
  - Tameside Hospital, Manchester
  - Whiston Hospital, Whiston

IPD SHARING:
Plan to Share IPD: Undecided
The current data sharing plans for this study are unknown and will be available at a later date